CLINICAL TRIAL: NCT04627519
Title: A Multicenter, Randomized, Open-label, Controlled Trial to Assess Effectiveness and Safety of Rhea Health Tone® as add-on Therapy for COVID-19 in Hospitalized Adults in Indonesia
Brief Title: Effectiveness and Safety of Rhea Health Tone® as add-on Therapy for COVID-19 in Hospitalized Adults in Indonesia
Acronym: RHEA-COVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitas Padjadjaran (Other)
Collaborators: PT. Rhea Pharmaceutical Sciences Indonesia (Unknown); Prodia Diacro Laboratories P.T. (Industry)
Responsible Party: Principal Investigator, Keri Lestari, Prof. Dr. Keri Lestari, M.Si, S.Si, Apt., Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pharm-202010.01
Record Dates: First submitted 2020-11-10; First posted 2020-11-13 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Covid19; Rhea Health Tone
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to be in Arm 1 or Arm 2 using pre-defined randomisation list; 1:1 for each arm.
  Arm 1 receives Standard of Care (day 1 to 10) Arm 2 receives Standard of Care + Rhea Health Tone (day 1 to 10)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoC alone (No Intervention): Standard of Care alone (days 1 to 9)
- Rhea Health Tone® (Experimental): Rhea Health Tone® 2 ml twice daily after meal (every 12 hours) for 9 days to be provided together with Standard of Care.
  Interventions: Dietary Supplement: Rhea Health Tone®

INTERVENTIONS:
Dietary Supplement: Rhea Health Tone® — Rhea Health Tone® 2 ml twice daily after the meal (every 12 hours)
  Arms: Rhea Health Tone®

SUMMARY:
This is a multicenter, randomized, open-label, controlled trial to evaluate the effectiveness and safety of Rhea Health Tone® as add-on therapy in hospitalized adults with COVID-19.

The study is a multi-center trial that will be conducted in up to approximately 2 sites nationally. New sites may be added as needed after appropriate assessment. Interim monitoring will be conducted to evaluate the arms and for safety and effectiveness. Any change would be accompanied by updated sample size.

Subjects will be assessed while hospitalized. All subjects will undergo a series of laboratory (inflammatory biomarkers (IL-6, hs-CRP, IFNγ), SGOT, SGPT and Creatinine, conversion rate by PCR, QTc prolongation by ECG, chest X-ray), clinical (clinical assessment, vital sign, concomitant medication, other medical conditions) and safety assessment (serious adverse event).

Randomization will be performed 1:1 for each arm. Arm 1 = Standard of Care (SoC) alone, arm 2 = SoC + Rhea Health Tone®.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, controlled trial to evaluate the effectiveness and safety of Rhea Health Tone® in hospitalized adults with COVID-19 confirmed by PCR.

The study is a multi-center trial that will be conducted in up to approximately 2 sites nationally. Interim monitoring will be conducted to evaluate the arms and for safety and effectiveness. Any change would be accompanied by an updated sample size.

Eligible patients are male or female adults (age ≥ 18 years up to 50 years old) recently admitted as in-patients, with mild to moderate COVID-19 confirmed by positive PCR that fulfill the inclusion and exclusion criteria stated in the protocol. Laboratory assessment include SGOT, SGPT and Creatinine at screening. The subjects must sign their consent in writing electronically beforehand. Total subjects = 69.

Subjects with any of these conditions will be excluded:

* Any allergy to any composition of Rhea Health Tone;
* Pregnant and breast feeding;
* History and co-morbid of severe underlying disease where treatment and follow up is not likely to be beneficial to the patient based on physician judgement (e.g. retinopathy, cardiovascular disease (QTc > 500 mdet (narrow QRS); QTc ≥ 550 mdet (wide QRS)), heart arrythmia, uncontrolled diabetes mellitus, hypertension, chronic pulmonary disease, asthma, chronic kidney disease (Creatinine > 2x upper limit of normal), liver disease (SGOT/SGPT > 2x upper limit of normal), chronic neurological disease, or etc.). This includes people requiring care in designated supported living facilities and severe dementia;
* Possibility of being transferred to a non-study-hospital within 72 hours.
* History of autoimmune disease, cancer, HIV AIDS

Any suspected serious adverse event reaction is reported to CRO/Sponsor and EC within 24 hours, using patient's study ID.

During the study conduct, the study team shall keep all the relevant source documents and transcribe the data in case report form (CRF). The study team should also update study essential document (e.g. subject log, investigational product accountability log, etc.) and keep the copy captured by scan/camera for monitoring/audit/inspection purpose.

The study is expected to be finished in 2 months.

Standard of Care (SoC) treatment is based on COVID-19 Treatment Protocol (1st edition, 2020) published by Medical Associations (PDPI, PERKI, PAPDI, PERDATIN, IDAI).

Arm 1: SoC alone for 9 days Arm 2: SoC + Rhea Health Tone 2 ml twice a day after meal (every 12 hours) for 9 days.

It is anticipated that patients with COVID-19 will present to participating hospitals, and that no external recruitment efforts towards potential subjects are needed. Recruitment efforts may also include dissemination of information about this trial to other medical professionals/hospitals.

The Ethics Committee will approve the recruitment process and all materials prior to any recruitment to prospective subjects directly.

Screening will begin with a brief discussion with study staff. Some will be excluded based on demographic data and medical history (i.e., pregnant, < 18 years of age, severe COVID-19, etc.). Information about the study will be presented to potential subjects (or legally acceptable representative) and questions will be asked to determine potential eligibility. Screening procedures can begin only after informed consent is obtained.

To evaluate the effectiveness of Rhea Health Tone® in the therapy of mild to moderate hospitalized adults with confirmed COVID-19 based on length of stay in hospital (after subject received randomization code until subject discharge/death/recovered). Secondary parameters will be Incidence and duration of Oxygenation (days of oxygenation), incidence is defined as number of days from randomization until the subject received oxygenation, duration is defined as total days of the use of oxygenation; incidence of Ventilation (days to receiving ventilation).

Incidence is defined as number of days from randomization until the subject received ventilation; inflammatory biomarkers (IL-6, hs-CRP and IFNγ).

Analyses relate outcome to the randomly allocated treatment (e.g. intent-to-treat). The primary analyses assess any effects of treatment allocation on length of hospitalization, analyzing separately people who already at mild and moderate level at entry and by age. Interim analysis will be carried out after 50% subject enrolled. The results will be monitored by monitor assigned by the Sponsor to ensure subject well-being and safety as well as study integrity. The monitor will evaluate the study safety parameter after 50% subject enrolled in the study.

The main secondary analyses assess any effects of treatment allocation on:

1. Incidence and duration of Oxygenation (days of oxygenation, days of free oxygenation);
2. Incidence of Ventilation (days to receiving ventilation);
3. Inflammatory biomarkers (IL-6, hs-CRP , IFNγ );
4. Conversion rate from positive to negative by PCR result;
5. Percentage of improvement of patients' clinical
6. Percentage of improvement of patients based on chest X-ray; and
7. QTc prolongation by ECG.

Study related data will be recorded. All the data in the source documents shall be collected by the study team to be transcribed in the electronic case report form (eCRF). Once the document recorded, the electronic data will be automatically available for monitoring/audit/inspection purpose. All the electronic system used and data recording in the study must be conducted in compliance to Good Clinical Practice.

The investigator must assure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On CRFs or other documents submitted to the sponsor, subjects should not be identified by their names, but by an identification code. The investigator should keep a subject enrolment log showing codes, names and addresses. The investigator should maintain documents not for submission to Sponsor, e.g. subjects' written consent forms, in strict confidence.

The investigator shall ensure the quality control and quality assurance of the data generated during the study and how the data will be handled, including providing access to monitoring activities, audit and inspection and source documents which will be used in the study. Investigator will permit monitoring, audits and inspections by Sponsor/CRO, EC, and regulatory bodies.

All source records including electronic data (if any) will be stored in secured systems in accordance with institutional policies and locally applicable regulation. All the essential documents should be retained until at least 5 years after the study ended or based on the applicable regulatory requirements or based on the agreement with the funder.

The Drug Safety Monitoring Board (DSMB) is an Independent Data Monitoring Committee consisting of doctors who are experienced in clinical trials, statisticians, and other members who do not direct involvement with this study. The DSMB responsible for the ongoing review of a clinical trial and for making recommendations to the sponsor concerning the continuation, modification, and termination of the trial as it is being conducted. The DSMB will be the only committee that is allowed to review the confidential data in the study. The statistician will analyze the subject's security data and report to DSMB to be evaluated more closely. The key responsibilities of the DSMB are to ensure patient safety by routine review of overall safety data including all SAEs, SUSARs, all severe AEs and AEs leading to drug or study discontinuation and, where applicable, literature cases and information from Competent Authorities (CAs) and by judging the relevance of the events for patients' safety. The DSMB will review the results of data that has been analyzed in accordance with SAP and consider other evidence arising from other studies and will provide advice to the Trial Steering Committee (TSC) (the research committee and national coordinator) regarding the sustainability of this study. The DSMB may recommend the TSC to the recruitment or study termination or provide recommendations related to alternatives treatment (if any).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years to 50 years old, who recently admitted as in-patients and have not received any standard of care yet, with COVID-19 confirmed by PCR with mild to moderate symptoms.
2. Female subjects of child-bearing age agree to take effective contraceptive measures during the study until seven days of the last oral medication of study product;
3. Willing to receive a random assignment to any designated treatment group and not participating in another study at the same time;
4. Willing for not using any other immunomodulator or treatment that might bias the study
5. Patient willing to provide informed consent.

Exclusion Criteria:

1. Any allergy to any composition of Rhea Health Tone®;
2. Pregnant and breastfeeding;
3. History and co-morbid of severe underlying disease where treatment and follow up is not likely to be beneficial to the patient based on physician judgment (e.g. retinopathy, cardiovascular disease (QTc > 500 mdet (narrow QRS); QTc ≥ 550 mdet (wide QRS)), heart arrhythmia, uncontrolled diabetes mellitus, hypertension, chronic pulmonary disease, asthma, chronic kidney disease (Creatinine > 2x upper limit of normal), liver disease (SGOT/SGPT > 2x limit of normal), chronic neurological disease, or etc.). This includes people requiring care in designated supported living facilities and severe dementia;
4. Possibility of being transferred to a non-study-hospital within 72 hours.
5. History of autoimmune disease, cancer, HIV AIDS.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Length of stay | From the date of randomization until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  Total days the subjects were hospitalized

SECONDARY OUTCOMES:
Duration of oxygenation | From the date of randomization until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  Total days of oxygen supplementation
Duration of ventilation | From the date of randomization until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  Total days of receiving ventilation
PCR conversion | Will be examined at days 1st , 7th, and 10th.
  Total days of conversion rate from positive to negative by PCR result
Inflammatory biomarkers 1 | Will be examined at days 1st and 10th.
  IL-6 (pg/mL)
Inflammatory biomarkers 2 | Will be examined at days 1st and 10th.
  hs-CRP (mg/L)
Inflammatory biomarkers 3 | Will be examined at days 1st and 10th.
  IFNγ (pg/mL)
Percentage of improvement of subjects' clinical status | From the date of randomization until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  Daily measurement of temperature, heart rate, respiratory rate, blood pressure, oxygen saturation, capillary filling time >2 seconds
X-Ray | From the date of informed consent signed by subject, until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  Percentage of improvement of subjects based on chest X-ray

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Rumah Sakit Darurat Penanganan Covid-19 Wisma Atlet Kemayoran (RSDCWA), Jakarta, DKI Jakarta
  - Dr. Hasan Sadikin Central General Hospital, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509
- [Result] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093
- [Result] Swamy MK, Akhtar MS, Sinniah UR. Antimicrobial Properties of Plant Essential Oils against Human Pathogens and Their Mode of Action: An Updated Review. Evid Based Complement Alternat Med. 2016;2016:3012462. doi: 10.1155/2016/3012462. Epub 2016 Dec 20. PMID 28090211
- [Result] Yang L, Peng K, Zhao S, Zhao F, Chen L, Qiu F. 2-methyl-L-erythritol glycosides from Gardenia jasminoides. Fitoterapia. 2013 Sep;89:126-30. doi: 10.1016/j.fitote.2013.05.018. Epub 2013 May 31. PMID 23727470
- [Result] Zhang Y, Yao J, Qi X, Liu X, Lu X, Feng G. Geniposide demonstrates anti-inflammatory and antiviral activity against pandemic A/Jiangsu/1/2009 (H1N1) influenza virus infection in vitro and in vivo. Antivir Ther. 2017;22(7):599-611. doi: 10.3851/IMP3152. Epub 2017 Mar 8. PMID 28272019
- [Result] Wu S, Patel KB, Booth LJ, Metcalf JP, Lin HK, Wu W. Protective essential oil attenuates influenza virus infection: an in vitro study in MDCK cells. BMC Complement Altern Med. 2010 Nov 15;10:69. doi: 10.1186/1472-6882-10-69. PMID 21078173
- [Result] Su S, Hua Y, Wang Y, Gu W, Zhou W, Duan JA, Jiang H, Chen T, Tang Y. Evaluation of the anti-inflammatory and analgesic properties of individual and combined extracts from Commiphora myrrha, and Boswellia carterii. J Ethnopharmacol. 2012 Jan 31;139(2):649-56. doi: 10.1016/j.jep.2011.12.013. Epub 2011 Dec 13. PMID 22178177
- [Result] Tipton DA, Lyle B, Babich H, Dabbous MKh. In vitro cytotoxic and anti-inflammatory effects of myrrh oil on human gingival fibroblasts and epithelial cells. Toxicol In Vitro. 2003 Jun;17(3):301-10. doi: 10.1016/s0887-2333(03)00018-3. PMID 12781209
- [Result] Nomicos EY. Myrrh: medical marvel or myth of the Magi? Holist Nurs Pract. 2007 Nov-Dec;21(6):308-23. doi: 10.1097/01.HNP.0000298616.32846.34. PMID 17978635
- [Result] Sharopov F, Valiev A, Satyal P, Gulmurodov I, Yusufi S, Setzer WN, Wink M. Cytotoxicity of the Essential Oil of Fennel (Foeniculum vulgare) from Tajikistan. Foods. 2017 Aug 28;6(9):73. doi: 10.3390/foods6090073. PMID 28846628
- [Result] Lee HS, Kang P, Kim KY, Seol GH. Foeniculum vulgare Mill. Protects against Lipopolysaccharide-induced Acute Lung Injury in Mice through ERK-dependent NF-kappaB Activation. Korean J Physiol Pharmacol. 2015 Mar;19(2):183-9. doi: 10.4196/kjpp.2015.19.2.183. Epub 2015 Feb 25. PMID 25729281
- [Result] Shalaby NM, Maghraby AS, el-Hagrassy AM. Effect of Daucus carota var. boissieri extracts on immune response of Schistosoma mansoni infected mice. Folia Microbiol (Praha). 1999;44(4):441-8. doi: 10.1007/BF02903720. PMID 10983240
- [Result] Alves-Silva JM, Zuzarte M, Goncalves MJ, Cavaleiro C, Cruz MT, Cardoso SM, Salgueiro L. New Claims for Wild Carrot (Daucus carota subsp. carota) Essential Oil. Evid Based Complement Alternat Med. 2016;2016:9045196. doi: 10.1155/2016/9045196. Epub 2016 Feb 14. PMID 26981143
- [Result] Yuan H, Ma Q, Cui H, Liu G, Zhao X, Li W, Piao G. How Can Synergism of Traditional Medicines Benefit from Network Pharmacology? Molecules. 2017 Jul 7;22(7):1135. doi: 10.3390/molecules22071135. PMID 28686181
- See also: Coronavirus — https://www.who.int/health-topics/coronavirus#tab=tab_1
- See also: Burhan E, Susanto A, Nasution S, Ginanjar E, Pitoyo C, Susilo A, et al. PROTOKOL TATALAKSANA COVID-19. 1st ed. Jakarta: Perhimpunan Dokter Paru Indonesia (PDPI); 2020. — https://ocw.ui.ac.id/pluginfile.php/2518/mod_resource/content/9/Versi%20Cetak%20Protokol%20Tatalaksana%20COVID-19-ok.pdf
- See also: Pranita E. Sembuh dari Covid-19, Menurut WHO ini Rerata Waktu Penyembuhan Corona [Internet]. 2020 — https://www.kompas.com/sains/read/2020/04/02/170300223/sembuh-dari-covid-19-menurut-who-ini-rerata-waktu-penyembuhan-corona?page=all
- See also: Al-Samarrai O, Hameed R, Naji N. Studying of Phytochemical, Nutritive values and Antioxidant ability of Commiphora myrrha. Al-Mustansiriyh J Pharm Sciences. 2017;17(1):52-63. — http://ajps.uomustansiriyah.edu.iq/index.php/AJPS/article/view/59
- See also: Phatak RS. Phytochemistry, Pharmacological Activities and Intellectual Property Landscape of Gardenia jasminoides Ellis: a Review. Pharmacogn J. 2015 Jul 8;7(5):254-65. — http://www.phcogj.com/sites/default/files/10.5530pj.2015.5.1.pdf
- See also: urishi Y, Hamidi A, Zargar M, Singh S, Saxena A. Potential role of natural molecules in health and disease: Importance of boswellic acid. J Med Plants Res. 2010;4(2):2778-85. — https://academicjournals.org/journal/JMPR/article-abstract/68BFC7723000
- See also: Imamu X, Yili A, Aisa HA, Maksimov VV, Veshkurova ON, Salikhov ShI. Chemical composition and antimicrobial activity of essential oil from Daucus carota sativa seeds. Chem Nat Compd. 2007 Jul;43(4):495-6. — https://link.springer.com/article/10.1007/s10600-007-0174-2
- See also: Shebaby WN. Evaluation of antioxidant, anticancer and immunomodulatory activities of wild carrot (Daucus carota ssp. carota) oil and its fractions. [Disertation]. University of Surrey; 2014. — http://epubs.surrey.ac.uk/856520/
- See also: Djilani A, Ducko A. The Therapeutic Benefits of Essential Oils. Nutrition, Well-Being and Health — https://www.intechopen.com/books/nutrition-well-being-and-health/the-therapeutic-benefits-of-essential-oils
- See also: ha R, Babikian Y, Babikian H, Khoa L, Wisoyo D, Srisombat S, et al. Efficacy of Natural Herbal Formulation against Acute Hepatopancreatic Necrosis Disease (AHPND) causing Vibrio parahaemolyticus in Penaeus vannamei — https://openventio.org/efficacy-of-natural-herbal-formulation-against-acute-hepatopancreatic-necrosis-disease-ahpnd-causing-vibrio-parahaemolyticus-in-penaeus-vannamei/
- See also: Jha R, Babikian Y, Babikian H, Wisoyo S, Asih Y, Srisombat S, et al. Effectiveness of Natural Herbal Oil Formulation against White Spot Syndrome Virus in Penaeus vannamei. J Pharmacogn Nat Prod — https://www.hilarispublisher.com/open-access/effectiveness-of-natural-herbal-oil-formulation-against-white-spotsyndrome-virus-in-penaeus-vannamei-2472-0992-1000123.pdf
- See also: Al-Jameel WH, Al-Mahmood SS. Similarities and differences of COVID-19 and avian infectious bronchitis from molecular pathologist and poultry specialist view point. Iraqi Journal of Veterinary Sciences. 2020 May 15; — https://vetmedmosul.com/article_164760.html
- See also: Nadjib B.M. Effective Antiviral Activity of Essential Oils and their Characteristic Terpenes against Coronaviruses: An Update. Journal of Pharmacology & Clinical Toxicology. 2020;8(1): 1138(19 March 2020) — http://www.jscimedcentral.com/Pharmacology/pharmacology-8-1138.pdf
- See also: Maggo S. Dhull P, Dubey AP, Brashier, et. al. Cytokine Storm Syndrome in COVID-19: Diagnosis and Management Strategies. International Journal of Health Sciences and Research [Internet]. 2020 May;10(5) — https://www.ijhsr.org/IJHSR_Vol.10_Issue.5_May2020/25.pdf